CLINICAL TRIAL: NCT02511860
Title: Burdock and Blood Pressure in African-American Women: A Randomized Controlled Trial
Brief Title: Burdock and Blood Pressure in African-American Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Proactive Health Labs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00000001
Record Dates: First submitted 2015-07-15; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — burdock complex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will consume a placebo pill containing methylcellulose.
  Interventions: Dietary Supplement: Placebo
- Active (Active Comparator): Patients will consume 850 mg of burdock twice per day.
  Interventions: Dietary Supplement: Burdock

INTERVENTIONS:
Dietary Supplement: Burdock — Subjects will consume burdock daily and will undergo laboratory tests to determine the effect of burdock, if any, on organ function.
  Other Names: Arctium lappa
  Arms: Active
Dietary Supplement: Placebo — Methylcellulose (inert) tablet taken as placebo
  Arms: Placebo

SUMMARY:
This is a study of women aged 18-65, to determine the physiological effects of consuming burdock root in supplement form. Burdock has long been used by herbalists for its diuretic and blood sugar lowering properties.

DETAILED DESCRIPTION:
This study will allow us to determine the effect of burdock consumption on basic laboratory tests such as the complete metabolic panel (CMP) as well as the effect on blood pressure over time. Participants will self-monitor their blood pressures and undergo lab testing. They will also complete symptom inventories to determine subjective factors that change with burdock consumption, such as menstrual water retention. Subjects will undergo electronic body composition testing before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to swallow tablets
* African-American race
* Able to travel to our clinic in Santa Monica

Exclusion Criteria:

* Severely low blood pressure
* Hypoglycemia
* Baseline creatinine over 1.2

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 6 weeks

SECONDARY OUTCOMES:
Body fat percentage | 6 Weeks
Extracellular/Total Body Water Ratio | 6 Weeks
Hemoglobin A1c | 6 weeks
Blood urea nitrogen | 6 weeks
Creatinine | 6 weeks
Fasting Blood Glucose | 6 weeks
Liver function tests | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. De, Principal Investigator — Proactive Health Labs